CLINICAL TRIAL: NCT02534831
Title: The Effect of Soft Tissue Manual Therapy Intervention on Lung Function in Severe Chronic Obstructive Pulmonary Disease: a Proof of Concept Study
Brief Title: Manual Therapy in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Rodrigo Torres, Rodrigo Torres-Castro, University of Chile
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KIN2012-1
Record Dates: First submitted 2015-08-26; First posted 2015-08-28 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Soft Tissue Manual Therapy Protocol (Experimental): Soft tissue manual therapy protocol. Seven techniques of manual therapy in 30 minutes.
  Interventions: Procedure: Soft tissue manual therapy protocol

INTERVENTIONS:
Procedure: Soft tissue manual therapy protocol — The STMTP consisted of a pre-determined set of seven (7) soft tissue techniques delivered as part of a single treatment session lasting approximately 30 minutes. The techniques and their respective durations were: suboccipital release (5 minutes), anterior thoracic myofascial and sternum release (5 minutes), anterior cervical myofascial release (5 minutes), costal ligament balance (5 minutes) and muscular energy technique (MET) to the following muscles - scalenes (1 minute and 40 seconds), pectoralis minor (1 minute and 40 seconds) and latissimus dorsi and serratus anterior (1 minute and 40 seconds)

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common preventable and treatable disease characterized by progressive airflow limitation that is associated with an inflammatory response to noxious particles or gases.

Manual therapy (MT) has been defined as a therapeutic intervention that uses the hands to provide treatment to the musculoskeletal and/or visceral systems. It includes techniques such as massage, myofascial release, muscle energy technique, ligament balance, joint mobilization and joint manipulation. The suggestion that MT could deliver long-term benefits to people with COPD was first put forward in 2009. Since then a number of small studies have reported medium term improvements in lung function and exercise capacity following repeated applications of MT intervention.

Our aim is to measure the immediate effect on lung function of a single application of soft tissue manual therapy in patients with severe and very-severe chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a common preventable and treatable disease characterized by progressive airflow limitation that is associated with an inflammatory response to noxious particles or gases.

Changes in the anatomy of the airways and lung parenchyma occur as the result of bronchial hypersecretion and bronchoalveolar instability which cause expiratory flow limitation and air trapping. This is known clinically as dynamic hyperinflation. The phenomenon leads to an increase in expiratory reserve volume, residual volume and functional residual capacity, also referred to as end expiratory lung volume. These increases limit tidal volume and inspiratory reserve volume eventually affecting inspiratory capacity. They alter the position of the ribs causing a state similar to sustained inspiration over time, often referred to as 'inspiratory block'. This phenomenon is responsible for the characteristic 'barrel chest' commonly seen in patients with more advanced stages of COPD. In this state the position of the diaphragm is flattened and shortened reducing its ability to generate force. Accessory respiratory muscles are recruited as a compensatory adaptation leading to shortening and over-activation of these muscles over time (over-adaptation). The surrounding cervicothoracic fascia contracts producing postural changes such as anterior projection of the head, neck hyperextension, increased thoracic kyphosis and internal rotation of shoulders. These changes contribute to an increase in chest tightness, a decrease in the ability to generate inspiratory pressures and volumes and an increase in the amount of effort required to breath.

Manual therapy (MT) has been defined as a therapeutic intervention that uses the hands to provide treatment to the musculoskeletal and/or visceral systems. It includes techniques such as massage, myofascial release, muscle energy technique, ligament balance, joint mobilization and joint manipulation. The suggestion that MT could deliver long-term benefits to people with COPD was first put forward in 2009. Since then a number of small studies have reported medium term improvements in lung function and exercise capacity following repeated applications of MT intervention.

Our aim is to measure the immediate effect on lung function of a single application of soft tissue manual therapy in patients with severe and very-severe chronic obstructive pulmonary disease.

We recruitment patients with COPD in Rehabilitation Program in Hospital San José de Santiago de Chile, and we assessment: total lung capacity (TLC); vital capacity (VC); residual volume (RV); expiratory reserve volume (ERV); inspiratory capacity (IC); and airway resistance (Raw). Secondary: heart rate (HR); respiratory rate (RR); and oxygen saturation (SpO2).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe or very severe COPD (GOLD: Stage III or IV)
* Medically stable with no exacerbations in the preceding two months

Exclusion Criteria:

* A rheumatoid condition
* Neuromuscular or musculoskeletal pathology
* Cognitive disability that could influence their understanding or execution of the assessment tests or intervention protocol
* Supplemental oxygen dependency
* Previous or current enrollment in other pulmonary rehabilitation program

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Total Lung Capacity | 30 minutes
  Units in ml

SECONDARY OUTCOMES:
Vital Capacity | 30 minutes
  Units in ml
Residual volume | 30 minutes
  units in ml

CONTACTS AND LOCATIONS:
Overall Officials: Roger Engel, PhD, Study Director — Macquarie University, Australia
Locations (1):
- Department of Physical Therapy, University of Chile, Santiago, Metropolitan Región, Chile